CLINICAL TRIAL: NCT00921609
Title: A Study Examining the Peri- and Post-operative Dynamics of the GH-IGF-1 Axis in Subjects With Acromegaly During the First Year After Surgical Resection
Brief Title: Peri-operative Dynamics of the Growth Hormone Axis in Subjects With Acromegaly
Status: Active, not recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Odelia Cooper, Associate Professor of Medicine, Division of Endocrinology, Diabetes, and Metabolism, Cedars-Sinai Medical Center
Other Study IDs: 8997
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Acromegaly
Keywords: Acromegaly; OGTT; post-op
MeSH Terms: conditions — Acromegaly | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1 ml frozen serum saved to run free IGF-1

GROUPS / COHORTS (1):
- Acromegaly patients: All patients will undergo oral glucose tolerance test at postoperative day 1, 6 weeks, 3 months, and 1 year
  Interventions: Diagnostic Test: Oral glucose tolerance test

INTERVENTIONS:
Diagnostic Test: Oral glucose tolerance test — An oral glucose tolerance test is a test that lowers growth hormone in the body to very low levels for a short time in order to see how low the growth hormone levels are in your blood.

SUMMARY:
Acromegaly is a rare disorder characterized by excessive production of growth hormone most often by a pituitary adenoma. A pituitary adenoma is a tumor, almost always benign or non-cancerous, that grows on the pituitary, a small gland located at the base of the brain. Treatment of acromegaly usually involves surgery, medication, or radiation, but can involve a combination of these three treatments.

Subjects for this study will be recruited if they are:

1. Adults, male or female, between the ages of 18-90.
2. Have been diagnosed with acromegaly, based on elevated levels of growth hormone, IGF-I (a hormone made in response to growth hormone), and a pituitary adenoma visualized on an MRI.
3. Patients would have already agreed to have their acromegaly treated with surgery prior to study entry.

Subjects will have measurements of growth hormone using an oral glucose tolerance test (OGTT), IGF-I, free IGF-I and levels of IGF binding proteins at four time points after their pituitary surgery: Day 1, Day 42 (6 weeks), Day 84 (12 weeks), and day 365 (1 year). Subjects will also have an MRI of the pituitary done at 12 weeks and 1 year. OGTT and IGF-I are routinely measured to assess whether or not a person is cured of their acromegaly. An MRI of the pituitary is routinely done at 12 weeks and 1 year after surgery to assess the results of surgery. Free IGF-I and IGF binding proteins are not routinely measured after surgery, but are being done to see if they relate more strongly to disease activity than IGF-I and growth hormone.

OGTT and the IGF-I binding proteins are not routinely measured on the day after surgery, but are being done to examine the predictive ability of these tests at a very early time after surgery. Data obtained from these tests will be compared to the data gathered at the 1 year time point.

IGF-I and growth hormone will be measured by a commercial clinical lab, Quest Diagnostics, for clinical decision-making at the time of service. IGF-I and growth hormone will also be measured using other methods to attempt to investigate the variability of these hormones when different assays are used.

DETAILED DESCRIPTION:
Acromegaly Overview

Acromegaly is a rare, insidious disorder characterized by excessive secretion of growth hormone (GH) almost always from a pituitary adenoma. (Melmed NEJM 1990) Excess GH secretion in turn leads to increased levels of insulin-like growth factor-I (IGF-I), which is primarily responsible for the clinical manifestations of the disease. Features of acromegaly are numerous and include acral and soft tissue growth, arthropathy, excessive sweating, glucose intolerance, and carpal tunnel syndrome. Many patients have cardiomyopathy and hypertension and the diagnosis of acromegaly carries with it an excessive morbidity and mortality related to cardiovascular disease.

Therapy

The goals of therapy include management of the pituitary mass, control of symptoms of GH excess, improvement in long term morbidity and mortality associated with GH excess, and biochemical normalization of IGF-I and GH secretion without disruption of normal anterior pituitary function. Treatment for acromegaly has generally included one or a combination of three modalities, surgery, radiation and medication.

Classically, surgery has been the primary treatment modality with surgical cure being dependent upon pituitary tumor size and the surgical expertise of the surgeon. In experienced hands, transsphenoidal surgical resection of pituitary adenomas is a low risk procedure with few peri-operative or long term complications. Published cure rates for microadenomas and macroadenomas range from 39-91% and 12-71%, respectively. (Melmed S, Kleinberg DL, Williams Textbook of Endocrinology.) Subjects who are not controlled with surgery alone require additional therapy in the form of radiation or medication.

Medical therapy is the preferred choice of second line therapies and is available in multiple forms including short and long acting somatostatin analog therapy aimed at reducing GH secretion via the SSTR2 receptor, dopamine agonist therapy (effective in only about 10% of patients) and pegvisomant, a GH receptor antagonist which lowers IGF-I levels but does not decrease GH secretion or control tumor size.

Radiation therapy is available in multiple modalities and is an effective form of controlling excessive GH secretion and tumor size. One drawback to radiation therapy is the length of time needed for the therapy to take effect. GH secretion gradually declines over several years and medical therapy is often needed to control GH secretion until radiation therapy has taken effect. The major side effect of all forms of radiation therapy is hypopituitarism, with approximately 50% of all subjects experiencing some form of hypopituitarism at 10 years.

Assessing Control

Since there is no well-defined clinical outcome to help establish if a patient is cured, the assessment of disease activity has generally relied on arbitrary biochemical parameters. These parameters include normalization of IGF-I when compared to age and gender matched normal values and reducing the GH response to glucose suppression to less than 1mcg/L. The level of GH suppression has evolved to the current level due to advances in the sensitivity of the growth hormone assay. Previous values of greater than 1mcg/L were based on the use of a less sensitive polyclonal radio-immunoassay (RIA) and have become obsolete with the widespread use of far more sensitive monoclonal assays (chemiluminescent, immunoradiometric, or immunoflourometric). Future improvements in GH assay sensitivity may alter the currently held cutoff point of 1mcg/L to even lower levels, but the clinical significance of these lower levels has yet to be established.

The amount of glucose used for the suppression of GH during an oral glucose tolerance test (OGTT) has been either 75g or 100g, and there has been no data establishing the superiority of one dose compared to the other. Recent consensus guidelines suggest the use of 75g of oral glucose for the purposes of standardization (Giustina et al, 2000, JCEM, Vol 85: p526-9).

Long-Term Management

Long-term follow-up of subjects treated for their acromegaly has shown an improvement in morbidity and mortality. Swearingen et al. (JCEM 1998 Vol. 83: p 3419-3426) showed that patient-years with persistence of disease, as defined by normalization of IGF-I, carried with it a 3.5 fold relative mortality risk compared to patient-years in remission using a Cox proportional hazards model. They were also able to demonstrate that subjects who had achieved control of their acromegaly showed similar survival rates to those in the general U.S. population. These data underscore the benefits of achieving control of acromegaly and draws attention to the need for accurate criteria for defining control and standardized methodology of observation following treatment of acromegaly.

GH-IGF-I Discordance and the Risk For Recurrence

Other investigators (Freda et al, 2004, JCEM 89: 495-500) have found that some post-operative subjects with acromegaly with normal IGF-I levels (age and gender matched) have persistently abnormal nadir GH responses to OGTT (100g dextrose; nadir GH >0.14 mcg/L). These subjects had an increased rate of disease recurrence when followed longitudinally as compared to post-operative subjects with normal IGF-I and normal nadir GH responses to OGTT (GH < 0.14 mcg/L).

Abnormal GH responses to OGTT in the setting of normal IGF-I levels may not be reflective of a "lack of cure" in subjects status-post surgical treatment for acromegaly. These subjects may be secreting elevated amounts of GH due to a lack of inhibition by lower levels of IGF-I. IGF-I levels may be considered normal in comparison to control data for the age and gender matched populations; but may be either low for that particular individual, or lower than IGF-I levels seen prior to treatment for acromegaly. In this setting, the IGF-I level is considered low and the normal pituitary tissue responds by secreting excessive amounts of GH in the absence of IGF-I suppression.

Recent data regarding the feedback mechanism responsible for GH release from pituitary somatotroph cells supports what has long been theorized: that circulating levels of free IGF-I, and not IGF-I bound to the IGF binding protein complex, suppress secretion of GH (Chen JW et al., 2005, JCEM 90: 366-371.) Generally, measuring levels of free IGF-I has not added any significant clinical data to the assessment of GH secretion in the diagnosis or management of acromegaly. However, it has been suggested that in situations where there is discordant information regarding the GH suppression in response to oral glucose and the measurement of total IGF-I, that free IGF-I levels may be a better indicator of GH secretion and bioactivity (Frystyk J, 2004, GH and IGF-I Research, 14: 337-75 and Feelders RA, 2005, JCEM 90: 6480-6489.)

Hypothesis: Assessment of post-operative subjects with low-normal IGF-I but non-suppressed nadir GH levels will show normalization over time with lower, normal nadir levels of GH in response to OGTT. IGF-I levels could increase over time, but would still be considered normal as compared to age and gender matched normal levels in subjects who are considered "controlled." Rather than consider subjects with abnormal responses to OGTT in the setting of low-normal IGF-I as "not cured" and at a higher risk for recurrence, these subjects may be exhibiting compensatory elevation of GH in the absence of IGF-I suppression. Over time, subjects with non-suppressed GH responses to OGTT and low-normal IGF-I would have lower GH nadirs in response to OGTT and persistently normal (although possibly higher than the post-operative initial assessment) IGF-I levels. This setting would be contrary to the expected elevation of IGF-I above normal limits in the setting of excess GH secretion.

Objectives: The primary objective of this study will be to determine the natural course of acromegaly treated with surgery in subjects with non-suppressed GH nadir values and normal total IGF-I values. A second objective of the study will be to determine the reliability of GH nadir to OGTT, free IGF-I, total IGF-I, and IGF binding proteins on post-operative day 1 in predicting long-term cure outcomes in acromegaly. A third objective will be to determine inter-assay variability in the measurement of GH and IGF-I levels.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female age 18-90
* Diagnosed with acromegaly from a pituitary adenoma visualized by MRI, and with elevated IGF-1 levels compared to age and gender matched control values and nadir GH response to OGTT>1mg/L
* Having already agreed to undergo surgical resection of their pituitary adenoma prior to study entry
* Must provide informed consent

Exclusion Criteria:

* Inability to complete the protocol due to intercurrent medical or psychiatric illness
* Pregnant or breastfeeding
* Use of insulin
* Use of estrogen, progesterone, testosterone or thyroid hormone will be allowed as long as the dose is stable during the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrollment will include subjects diagnosed with acromegaly caused by GH secreting adenomas who undergo surgical treatment for their disease provided they meet all inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2006-06 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Correlation of normalization of Growth hormone postoperatively with 1 year remission rates | 1 year
  The primary endpoint will be to assess if a higher proportion of subjects in group 2b (low normal IGF-1 and elevated GH) normalize their GH nadir responses to OGTT than subjects in group 2a (high normal IGF-1 and elevated GH) at either the three month time point or 12 month time point.

SECONDARY OUTCOMES:
Predictor of remission | 1 year
  A second objective of the study will be to determine the reliability of GH nadir to OGTT, free IGF-I, total IGF-I, and IGF binding proteins on post-operative day 1 in predicting long-term cure outcomes in acromegaly.
Assay variability of IGF-1 and GH | 1 year
  A third objective will be to determine inter-assay variability in the measurement of GH and IGF-I levels.

CONTACTS AND LOCATIONS:
Overall Officials: Odelia Cooper, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Pituitary Center, Los Angeles, California, United States